CLINICAL TRIAL: NCT02200666
Title: Forxiga Tablets Specific Clinical Experience Investigation for Long-term Use
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1692C00014
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Diabetes; Forxiga; Long-term use
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the investigation is to confirm the following under the post-marketing actual use of Forxiga Tablets (hereinafter referred to as Forxiga)

* Development of ADRs specified as Key Investigation Items and the risk factors
* Contributing factors possibly having an impact on the safety and efficacy
* Development of ADRs unexpected from the Precautions for use and ADRs under actual drug use

ELIGIBILITY:
Inclusion Criteria:

Patients treated with Forxiga for the first time due to type 2 diabetes mellitus, which is the indication of the drug.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Forxiga for the first time due to type 2 diabetes mellitus, which is the indication of the drug.
Sampling Method: Non-Probability Sample
Enrollment: 7793 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | from baseline to 3 years

CONTACTS AND LOCATIONS:
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3067&filename=JP_PMS%20Protocol_FXG_D1692C00014_E_Redacted.pdf
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1692C00014&attachmentIdentifier=28022cf7-726c-4258-b5cc-d32639730783&fileName=CSR_synopsis_D1692C00014.pdf&versionIdentifier=